CLINICAL TRIAL: NCT06605170
Title: Translation, Cross-cultural Adaptation, Reliability and Validity of the Traumatic Injuries Distress Scale to Turkish
Brief Title: Reliability and Validity of the Traumatic Injuries Distress Scale to Turkish
Status: Completed | Type: Observational
Sponsor: Uludag University (Other)
Responsible Party: Principal Investigator, Selim Mahmut GÜNAY, Principal Investigator, Uludag University
Other Study IDs: 2020-13/21
Record Dates: First submitted 2024-09-12; First posted 2024-09-20 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Musculoskeletal Injury; Trauma Injury
Keywords: TIDS; Reliability; Validity; TIDS-TR
MeSH Terms: conditions — Accidental Injuries | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire — Translate and culturally adapt the original English version of the traumatic injuries distress scale to Turkish

SUMMARY:
The Traumatic Injuries distress Scale is a patient-reported measure that assesses suffering following non-catastrophic musculoskeletal injuries. The original English version demonstrated acceptable accuracy in predicting recovery trajectories up to 12 months later. This study aimed to determine the cultural adaptation, validity and reliability of the Turkish version of TIDS-TR in young and physically active patients with hip pain.

DETAILED DESCRIPTION:
The Traumatic Injuries distress Scale (TIDS) is commonly used to measure methods of coping with various forms of Traumatic Injuries. TIDS is a self-report questionnaire developed by David M. Walton et al. in 2016 to assess the magnitude of stress experienced as a result of recent musculoskeletal trauma. It is administered between 2 days and 4 weeks after injury and is used to estimate the likelihood of recovery within 6 to 12 months. Each item in the TIDS questionnaire, which consists of 12 items, is scored as 0, 1, or 2, and the total score is at least 0 and at most 24. The total TIDS score is interpreted as low risk (≤ 3), medium or unknown risk (4 to 10), and high risk (≥ 11) according to the score obtained. TIDS consists of three subscales: 1) uncontrolled pain (4 items), 2) negative affect (6 items), and 3) intrusion/hyperarousal (2 items). Each of the subscales has guiding features for clinicians to determine treatment priorities such as pain management, cognitive or psychological intervention, and stress management techniques. It is recommended that when the uncontrolled pain subscale score is 3 and above, the applications should be aimed at symptom control, when the negative affect score is 3 and above, the applications should be aimed at correcting negative mood, and when the intrusion/hyperarousal score is 1 and above, the applications should be aimed at treating anxiety and post-traumatic stress disorder.

The questionnaires validity and reliability were examined, and good findings were found, leading to the tools widespread use. The purpose of this study was to translate and culturally adapt the original English version of the TIDS into Turkish, as well as to evaluate the instruments validity and reliability in patients with traumatic musculoskeletal injury.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old,
* Having good reading and writing skills in Turkish,
* Having suffered a traumatic musculoskeletal injury that does not require surgery or inpatient treatment
* At least 2 and at most 4 weeks have passed since the injury

Exclusion Criteria:

* Those with organ disease
* Those with blood clotting disorders
* Those with neuromuscular disorders
* Those with rheumatoid diseases
* Those with cancer
* Those with systemic diseases such as uncontrollable psychopathology

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Those who have suffered traumatic musculoskeletal injuries that do not require surgery or inpatient treatment
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2024-09-30 (Actual); Primary Completion 2024-11-15 (Actual); Study Completion 2024-11-22 (Actual)

PRIMARY OUTCOMES:
Age of the patients | 4 weeks
  Age will be recorded.
Gender of the patients | 4 weeks
  Gender will be recorded.
body mass index of the patients | 4 weeks
  body mass index will be recorded.
education level of the patients | 4 weeks
  education level will be recorded.
employment status of the patients | 4 weeks
  employment status will be recorded.
duration of pain of the patients | 4 weeks
  duration of pain will be recorded.
duration, type and location of pain of the patients | 4 weeks
  duration, type and location of pain will be recorded.
type of injury of the patients | 4 weeks
  type of injury will be recorded.
mechanism of injury of the patients | 4 weeks
  mechanism of injury will be recorded.
Traumatic Injuries Distress Scale | 4 weeks
  Traumatic Injuries Distress Scale questionnaire will be filled out under the supervision of a physiotherapist.
Hospital Anxiety and Depression Scale (HADS) | 4 weeks
  Hospital Anxiety and Depression Scale (HADS) questionnaire will be filled out under the supervision of a physiotherapist.
Short Form-12 (SF-12) | 4 weeks
  Short Form-12 (SF-12) questionnaire will be filled out under the supervision of a physiotherapist.

CONTACTS AND LOCATIONS:
Overall Officials: Selim Mahmut GÜNAY, Dr, Study Chair — Uludağ University
Locations (1):
- Uludag University, Bursa, Nilüfer, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Walton DM, Krebs D, Moulden D, Wade P, Levesque L, Elliott J, MacDermid JC. The Traumatic Injuries Distress Scale: A New Tool That Quantifies Distress and Has Predictive Validity With Patient-Reported Outcomes. J Orthop Sports Phys Ther. 2016 Oct;46(10):920-928. doi: 10.2519/jospt.2016.6594. Epub 2016 Sep 3. PMID 27594662